CLINICAL TRIAL: NCT01794975
Title: Changes in Striatal [11C]ORM-13070 Binding Elicited by Changing Levels of Endogenous Noradrenaline - a PET Study in Healthy Human Subjects
Brief Title: Changes in Striatal [11C]ORM-13070 Binding Elicited by Changing Levels of Endogenous Noradrenaline
Acronym: AIMI2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Turku University Hospital (Other Government); Orion Corporation, Orion Pharma (Industry)
Responsible Party: Principal Investigator, Juha Rinne, Professor, MD, PhD, University of Turku
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: AIMI 2
Record Dates: First submitted 2013-02-15; First posted 2013-02-20 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Changes in Striatal [11C]ORM-13070 Binding.
Keywords: PET; striatum; receptor occupancy; noradrenaline; alpha2c
MeSH Terms: interventions — Ketamine; Atomoxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ketamine (Active Comparator): Ketamine will be administered intravenously using a pseudo steady state infusion approach with a target plasma concentration of 300 ng/ml starting 15 minutes before the PET scan and continued throughout the scan.
  Interventions: Drug: Ketamine; Drug: Placebo
- Atomoxetine and the cold pressor test (Active Comparator): An oral dose of approximately 1.2 mg/kg (range, 1.12-1.26 mg/kg) of atomoxetine is administered 1 h before the PET scans. A cold pressor test is employed as a physiological noradrenergic stimulus. The subject's foot is placed in a 8 °C water basin for the duration of the PET scan.
  Interventions: Drug: Atomoxetine; Other: Cold pressor test; Drug: Placebo
- Placebo (Placebo Comparator): Placebo capsules are given to mimic the atomoxetine treatment at each treatment visit except the atomoxetine visit. A baseline PET scan with [11C]ORM-13070 will be performed for all subjects with the placebo treatment only.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketamine
  Other Names: Ketalar
  Arms: Ketamine
Drug: Atomoxetine
  Other Names: Strattera
  Arms: Atomoxetine and the cold pressor test
Other: Cold pressor test
  Other Names: Cold stimulation of the subject's foot
  Arms: Atomoxetine and the cold pressor test
Drug: Placebo

SUMMARY:
The primary objective of the study is to further investigate whether striatal [11C]ORM-13070 uptake can be reduced by physiological and pharmacological challenges that increase the synaptic concentrations of noradrenaline in the human brain. Each subject will undergo 3 PET scans, a baseline PET scan and two scans with noradrenaline challenges: intravenous administration of ketamine and oral administration of atomoxetine combined with a cold pressor test where the subject's foot is placed in an 8 °C water basin. Eight healthy male subjects will be included in the study.

DETAILED DESCRIPTION:
Objectives

The primary objective of the study is to further investigate whether striatal [11C]ORM-13070 uptake can be reduced by physiological and pharmacological challenges that increase the synaptic concentrations of the endogenous alpha2C-adrenoceptor agonist, noradrenaline, in the human brain.

Methodology

PET will be used to study the effects of two different noradrenaline challenges on the striatal uptake of the novel alpha2C-adrenoceptor imaging agent, [11C]ORM-13070. Each of the eight study subjects will undergo one baseline PET scan without any pretreatment and two scans with two different noradrenaline challenges: i.v. infusion of ketamine and a single oral dose of atomoxetine combined with cold pressor test. The sequence of the baseline scan and the other scans for each subject will be based on balanced randomization. Double-blind administration of the pretreatments will not be possible, but the PET scanning data will be analyzed by a person who is not aware of the treatment identity. Venous blood samples will be collected for determination of concentrations of the [11C]ORM-13070 tracer and its radioactive metabolites, the test drugs atomoxetine and ketamine, and endogenous noradrenaline as a biomarker of the employed challenges. Blood pressure and heart rate will be measured as physiological indicators of sympathetic activation. Subject safety will be monitored by vital signs, questioning and clinical observation. The binding potential of the tracer in the striatum at baseline will be compared with the tracer binding potential after each of the noradrenaline challenges.

Sample size

Eight healthy male subjects will be included in the study. Discontinued subjects may be replaced by new subjects as decided by the Principal Investigator

Duration of treatment

After the screening visit, there will be an interval of no more than 45 days before the first PET visit. Each subject will undergo 3 PET scans: a baseline PET scan, and two scans with noradrenaline challenges. The PET experiments of each subject will be separated by intervals of at least 5 days. An end-of-study visit will take place within 21 days after the last PET scan.

Assessments

Efficacy: Alpha2C-adrenoceptor occupancy in the caudate nucleus and putamen will be assessed using the PET imaging agent [11C]ORM-13070 after the administration of two noradrenaline challenges, ketamine and atomoxetine combined with the cold pressor test. Differences in striatal receptor occupancy of the tracer will be assessed using established reference tissue models and the binding potentials of the non-displaceable compartment (BPND) according to the equation: Occupancy = [(BPND bl - BPND challenge) / BPNDbl x 100%]. Plasma noradrenaline concentrations will be measured as a biochemical biomarker before and after the interventions to validate the employed noradrenaline challenges. Blood pressure and heart rate will be used as physiological biomarkers.

Safety: Vital signs, subjective symptoms and ECG will be monitored during the PET visits. Subjects will remain at the study center for a minimum of 4 h after each PET scan, after which the subject will be discharged based on clinical evaluation with a safety check list.

Pharmacokinetics: Venous blood samples will be collected for determination of concentrations of the [11C]ORM-13070 tracer and its radioactive metabolites, and the pretreatment agents atomoxetine and ketamine at pre-defined time points in order to provide information on the fraction of intact tracer in blood and to document the exposure to the pharmacological agents during the PET scans. No formal pharmacokinetic calculations will be performed.

Statistical methods:

Efficacy, safety and pharmacokinetics: Differences in striatal [11C]ORM-13070 uptake between the baseline condition and the different pretreatments will be considered a primary outcome variable and statistical analysis will be carried out with analysis of variance. Descriptive statistical analysis of the tracer fractions in blood during the scans and the concentrations of the employed pretreatment agents will be carried out. Demographic and other baseline data, laboratory safety determinations, physical examination, BP, HR, ECG, AEs and concomitant treatments will be summarised with descriptive statistics or listed.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent (IC) obtained.
2. Good general health ascertained by detailed medical history, laboratory investigations and physical examination.
3. Males between 20 and 40 years of age (inclusive).
4. Body mass index (BMI) between 18-28 kg/m2 (inclusive).
5. Weight 60-100 kg (inclusive).

Exclusion Criteria:

1. Suspected poor compliance with the protocol or inability to communicate well with the study personnel.
2. Veins unsuitable for repeated venipuncture.
3. CYP2D6 slow metabolizer or ultrarapid metabolizer genotype.
4. Evidence of clinically significant cardiovascular, renal, hepatic, haematological, gastrointestinal, pulmonary, metabolic-endocrine, neurological, urogenital or psychiatric disease as judged by the investigator.
5. Any condition requiring regular concomitant medication including herbal products or likely to need any concomitant medication during the study.
6. Susceptibility to severe allergic reactions.
7. Intake of any medication that could affect the outcome of the study, within 2 weeks prior to the tracer administration (2 months for enzyme inducing drugs like rifampicin or carbamazepine), or less than 5 times the half-life of the medication.
8. Regular consumption of more than 21 units of alcohol per week (1 unit = 4 cl spirits, about 13 g of alcohol).
9. Current use of nicotine-containing products more than 5 cigarettes or equivalent/day.
10. Inability to refrain from using nicotine-containing products during the stay at the study centre.
11. Inability to refrain from consuming caffeine-containing beverages during the stay at the study centre, e.g. propensity for headache when refraining from caffeine-containing beverages.
12. Blood donation or loss of significant amount of blood within 2 months prior to the screening visit.
13. Abnormal 12-lead electrocardiogram (ECG) finding of clinical relevance after 10 minutes rest in supine position at the screening visit
14. Heart rate (HR) < 40 beats/minute or > 90 beats/minute after 10 minutes rest in supine position at the screening visit.
15. At the screening visit, systolic blood pressure (BP) < 90 mmHg or > 140 mmHg after 10 minutes in supine position, diastolic BP < 50 mmHg or > 90 mmHg after 10 minutes in supine position.
16. Any abnormal laboratory value, vital sign or physical examination result, which may in the opinion of the investigator interfere with the interpretation of the test results or cause a health risk to the subject if he takes part in the study.
17. History of drug abuse or positive result in drug abuse test.
18. Positive serology to human immunodeficiency virus antibodies (HIVAb), hepatitis B surface antigen (HBsAg) or hepatitis C virus antibodies (HCVAb).
19. Anatomical abnormality in brain MRI which may in the opinion of the investigator interfere with the interpretation of the PET results.
20. Any other condition that in the opinion of the investigator would interfere with the evaluation of the results or constitute a health risk to the subject.
21. Participation in another clinical drug study within 3 months prior to this study.
22. Participation in a prior PET study or other medical or occupational exposure to significant doses of ionizing radiation.
23. Any contraindication to MRI of the brain.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2012-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Receptor occupancy | 5-30 minutes
  Alpha2C-adrenoceptor occupancy in the striatum will be assessed by comparing the amount of tracer uptake during the control scan to the amount of tracer uptake during the noradrenaline challenges. This assessment will be made once the results of all 3 scans are available for each subject.

CONTACTS AND LOCATIONS:
Overall Officials: Juha Rinne, PhD, Principal Investigator — Turku PET Centre
Locations (1):
- Clinical Research Services Turku (CRST) / Turku PET Centre, Turku, Finland